CLINICAL TRIAL: NCT01943071
Title: Effects and Costs of a Day Care Centre Program Designed for People With Dementia - a 24 Month Controlled Study
Brief Title: Effects and Costs of a Day Care Centre Program Designed for People With Dementia
Acronym: ECOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCAH-ECOD
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Dementia
Keywords: dementia; day care centre programs; patients; family carers; cost-consequence analysis
MeSH Terms: conditions — Dementia | interventions — Day Care, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Day care for patients with dementia (Experimental): Day care for patients with dementia
  Interventions: Behavioral: Day care for patients with dementia
- Care as usual (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Day care for patients with dementia — Day care centres designed by the local authorities for patients with dementia
  Arms: Day care for patients with dementia

SUMMARY:
Attending day care centres with programs specifically designed for patients with dementia is believed to postpone admittance to nursing home as well as increase quality of life and well-being for both patients and their family caregivers. We aim to investigate to what degree attendance in day care centres with programs for people with dementia is effective for patient and their caregivers whilst also cost efficient for society. The study consists of a quasi-experimental trial with comparison group. 400 patients with dementia, along with a family caregiver, will be included in the trial. Effects will be measured at baseline, after one and two years. Data collection will be made at three levels; at patient level with measures of cognition, depression, quality of life, functioning in activities in daily living, neuropsychiatric symptoms and death; at caregiver level with measures of depression, level of burden and quality of life; and at societal level with measures of nursing home admittance, hospital stays and use of other health resources. Additionally,a qualitative interview study will include 20 dyads from the main trial. The main focus will be on how attending day care centre programs for patients with dementia affect the lives of both patients and caregivers. Five of these dyads will be followed closely throughout the participation period to be used as case examples.

DETAILED DESCRIPTION:
A quasi experimental trial with a comparison group will be performed to evaluate the effect of the day care centre programs by comparing results from municipalities with (intervention group) and without (comparison group) a day care centre program designed for people with dementia using standardized assessment tools. Furthermore, a survey will be used to explore the communication and co-operation between the professional staff at the day care centre, the patients and the family carers by administering questionnaires to all three parties. Only patients with mild degree of dementia will be asked to participate in the questionnaire. Finally, qualitative interviews will be made with 20 dyads of patients and family carers to collect their in depth experience with the day care centre program. Five of these patients and their family carers will be followed closely as case examples for two years.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years or more and living at home
* Patients in the day care centre group must have attended the centre for at least four weeks and have been there no longer than nine months
* Dementia of either Alzheimer's type, vascular dementia, dementia with Lewy bodies/Parkinson's disease or a mixture of these types of dementias
* Capacity to give informed consent as judged by the professional caregivers
* A Mini Mental Status Examination (MMSE) score of ≥15
* Having a family carer willing to participate, who see the patients personally at least once a week
* Attending the day care centre program at least twice a week

Exclusion Criteria:

* Having applied for nursing home placement
* Suffering from a serious co-morbid physical disorder with life expectancy less than six months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 261 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Admittance to nursing home care | 24 months
  The number of patients admitted to nursing home care during a period of 24 months will be the primary outcome for the effect and the cost-consequence analysis

SECONDARY OUTCOMES:
Change in Quality of life for patients | 12 and 24 months
  The quality of life for patients as measured by Quality of Life - Alzheimer's Disease (QoL-AD)
Change in the patient's functioning of daily living | 12 and 24 months
  The Physical self-Maintenance Scale and Instrumental Activities of Daily Living Scale will be used to assess change in the patient's function of daily living
Change in depressive symptoms in patients | 12 and 24 months
  The change in depressive symptoms will be assessed by Montgomery Asberg Depression Rating Scale (MADRS)by interviews with both patient and family carer and the Cornell Scale for Depression in Dementia (CSDD) by interviews with family carers and a professional caregiver
Change in patient's cognition | 12 and 24 months
  Patient's cognition will be assessed using the Mini Mental State Examination (MMSE) the Clock Drawing Test (CDT), the Trail Making Test A (TMT-A)and the 10 word test of the Consortium to Establish a Registry in Alzheimer's Disease (CERAD)
Change in neuropsychiatric symptoms in patients | 12 and 24 months
  The change in Neuropsychiatric symptoms will be assessed using Neuropsychiatric Inventory Questionnaire (NPI-Q)
Patients death | 24 months
  Number of patients that have died during 24 months will be registered
Change in level of burden in family carers | 12 and 24 months
  Level of burden for family carers will be assessed by using the Relative's Stress Scale (RSS)
Change in family carers depressive symptoms | 12 and 24 months
  The MADRS will be used to assess depressive symptoms in family carers
Change in quality of life for family carers | 12 and 24 months
  QoL-AD will be used to assess quality of life in family carers
Differences in the use of health resources between the intervention group and the control group | 12 and 24 months
  The use of health resources will be measured using the resource Utilization in Dementia scale (RUD)
Differences in quality adjusted life years between the intervention group and the control group | 12 and 24 months
  A generic instrument, the EuroQol (EQ-5D) will be used to measure quality adjusted life years

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, Professor, Study Chair — Norwegian Centre for Ageling and health
Locations (1):
- Norwegian centre of Ageing and Health, Tønsberg, Norway

REFERENCES:
- [Derived] Rokstad AMM, Engedal K, Kirkevold O, Benth JS, Selbaek G. The impact of attending day care designed for home-dwelling people with dementia on nursing home admission: a 24-month controlled study. BMC Health Serv Res. 2018 Nov 16;18(1):864. doi: 10.1186/s12913-018-3686-5. PMID 30445937